CLINICAL TRIAL: NCT00617487
Title: Stress Echocardiography in the Early Identification of Pulmonary Arterial Hypertension in Systemic Sclerosis
Brief Title: Pulmonary Arterial Hypertension in Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Carlomaurizio Montecucco, Director, Dept. of Rheumatology, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: EchostressSSc
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Systemic Sclerosis; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Scleroderma, Systemic; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the role of stress echocardiography, compared to standard echocardiography in the early identification of pulmonary arterial hypertension in systemic sclerosis. To evaluate the role of BNP in this setting.To analyze data recorded with respect to the parameters commonly used for SSc evaluation (eg thorax HRCT, pulmonary function tests + DLCO, nailfold capillaroscopy, etc); these parameters are available starting for 1999.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic sclerosis according to LeRoy criteria

Exclusion Criteria:

* Pregnancy
* Significant valvular disease
* Low left ventricular function upon echocardiography (ejection fraction<55%)
* History of atrial fibrillation, myocardial infarction, pulmonary thromboembolisms, neoplasia or severe hepatic disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with systemic sclerosis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-12; Primary Completion 2018-03 (Estimated); Study Completion 2020-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Ghio, MD, Study Director — IRCCS Foundation Policlinico S. Matteo, Cardiology; Lorenzo Cavagna, MD, Principal Investigator — University and IRCCS Foundation Policlinico S. Matteo, Rheumatology
Locations (2):
- Italy (2):
  - IRCCS Foundation Policlinico S. Matteo, Pavia, PV
  - IRCCS Policlinico S. Matteo, Pavia, PV

REFERENCES:
- [Derived] Cavagna L, Caporali R, Klersy C, Ghio S, Albertini R, Scelsi L, Moratti R, Bonino C, Montecucco C. Comparison of brain natriuretic peptide (BNP) and NT-proBNP in screening for pulmonary arterial hypertension in patients with systemic sclerosis. J Rheumatol. 2010 Oct;37(10):2064-70. doi: 10.3899/jrheum.090997. Epub 2010 Jul 15. PMID 20634241